CLINICAL TRIAL: NCT01743560
Title: A Phase IV Multicentre, Open Label Study of Postmenopausal Women With Oestrogen Receptor Positive Locally Advanced or Metastatic Breast Cancer Treated With Everolimus (RAD001) in Combination With Exemestane, With Exploratory Epigenetic Marker Analysis
Brief Title: An Open Label Study of Postmenopausal Women With Oestrogen Receptor Positive Locally Advanced or Metastatic Breast Cancer Treated With Everolimus (RAD001) With Exemestane, With Exploratory Epigenetic Marker Analysis
Acronym: 4EVERUK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001YGB11; 2012-003689-41 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-12-06 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Oestrogen Receptor Positive Advanced Breast Cancer
Keywords: Breast Neoplasms; Neoplasms; Breast diseases; Skin diseases; Exemestane; Antibiotics, Antineoplastic; Everolimus; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions; Immunosuppressive Agents; Physiological Effects of Drugs; Aromatase Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Breast Diseases; Skin Diseases | interventions — Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus and Exemestane (Experimental): Postmenopausal women diagnosed with oestrogen receptor positive locally advanced or metastatic breast cancer will receive RAD001 at a dose of 10mg daily p.o. and exemestane 25mg daily p.o. for 48 weeks.
  Interventions: Drug: RAD001; Drug: Exemestane

INTERVENTIONS:
Drug: RAD001 — All postmenopausal women with oestrogen receptor positive locally advanced or metastatic breast cancer were treated with oral tablet RAD001 at a dose of 10mg daily and oral tablet exemestane 25mg daily. The study treatment for an individual patient was to begin on Study Day 1 and continue until the last patient enrolled completed the study at day 336 or until disease progression; unacceptable toxicity, death or early discontinuation from the study for any other reason, whichever occurs first.
  Other Names: Everolimus
Drug: Exemestane — All postmenopausal women with oestrogen receptor positive locally advanced or metastatic breast cancer were to be treated with oral tablet RAD001 at a dose of 10mg daily and oral tablet exemestane 25mg daily. The study treatment for an individual patient was to begin on Study Day 1 and continue until the last patient enrolled completed the study at day 336 or until disease progression; unacceptable toxicity, death or early discontinuation from the study for any other reason, whichever occurs first.

SUMMARY:
Determine the overall response rate (ORR) at 48 weeks to everolimus (RAD001, 10mg daily p.o.) and exemestane (25mg daily p.o.) treatment in postmenopausal women with oestrogen receptor positive breast cancer who have previous experienced recurrence or progression on non-steroidal aromatase inhibitor (NSAI) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of oestrogen receptor positive (ER+) and/or progesterone receptor positive (PgR+), human epidermal growth factor receptor 2 (HER2) negative breast cancer.
* Availability of archival tumour tissue (the tissue block or slides will be sent to the central laboratory for analysis).
* Postmenopausal women. The investigator must confirm postmenopausal status. Postmenopausal status is defined either by:

  * Age ≥ 55 years and one year or more of amenorrhea
  * Age < 55 years and one year or more of amenorrhea and postmenopausal levels of FSH and LH per local institutional standards
  * Prior hysterectomy and has postmenopausal levels of Follicle stimulating hormone (FSH) and Luteinizing Hormone (LH) per local institutional standards Surgical menopause with bilateral oophorectomy
* Disease progression following prior therapy with NSAI, defined as:

  * Recurrence while on or after completion of an adjuvant treatment including letrozole or anastrozole, or
  * Progression while on or following the completion of letrozole or anastrozole treatment for locally advanced or metastatic breast cancer

Note: Non-steroidal aromatase inhibitors (i.e. letrozole or anastrozole) do not have to be the last treatment prior to enrollment. Other prior anticancer therapy, e.g. tamoxifen, fulvestrant, exemestane are also allowed. Patients must have recovered to grade 1 or better from any adverse events (except alopecia) related to previous therapy prior to enrollment.

- Radiological evidence of recurrence or progression on last systemic therapy prior to enrollment.

Patients must have:

* At least one lesion that can be accurately measured or
* Bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease

  - Adequate bone marrow and coagulation function as shown by:
* Absolute neutrophil count (ANC) ≥ 1.5 109/L
* Platelets ≥ 100 ×109/L
* Hemoglobin (Hb) ≥ 9.0 g/dL
* International Normalized Ratio (INR) ≤ 2 .

  - Adequate liver function as shown by:
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN (or ≤ 5 if hepatic metastases are present)
* Total serum bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for patients known to have Gilbert Syndrome)

  - Adequate renal function as shown by:
* Serum creatinine ≤ 1.5 × ULN

  * Fasting serum cholesterol ≤ 300 mg/dl or 7.75 mmol/L and fasting triglycerides ≤ 2.5 × ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy and when the above mentioned values have been achieved
  * Eastern Cooperative Oncology Group (ECOG) performance status of PS </ 2
  * Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion Criteria:

* HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
* Pre-menopausal, pregnant, lactating women.
* Known hypersensitivity to mammilian target of Rapamycin (mTOR) inhibitors, e.g. sirolimus (rapamycin) or to their excipients.
* Known hypersensitivity to exemestane, to the active substance or to any of the excipients.
* Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption.
* Radiotherapy within four weeks prior to enrollment except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to enrollment. Patients must have recovered from radiotherapy toxicities prior to enrollment.
* Currently receiving hormone replacement therapy, unless discontinued prior to enrollment.
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use, at the time of study entry except in cases outlined below:

Prolonged systemic corticosteroid treatment during study, except for topical applications (e.g. rash),inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) should not be given. However:

* short duration (<2 weeks) of systemic corticosteroids is allowed (e.g. chronic obstructive pulmonary disease, anti-emetic)
* low doses of corticosteroids for brain metastasis treatment is allowed
* Patients with symptomatic visceral metastasis (e.g. significant dyspnoea related to pulmonary lymphangitic carcinomatosis and lung metastases or clinically meaningful symptomatic liver metastasis)
* Symptomatic brain or other Central Nervous system (CNS) metastases.
* Active, bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin, low molecular weight heparin (LMWH) and acetylsalicylic acid or equivalent, as long as the INR is 2.0)
* Any severe and / or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to enrollment, serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN
  * Acute and chronic, active infectious disorders (except for Hep B and Hep C positive patients) and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome)
  * Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude restrictive pulmonary disease, pneumonitis or pulmonary infiltrates.
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (rifabutin, rifampicin, clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir, telithromycin) within the last 5 days prior to enrollment
* History of non-compliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Another malignancy within 5 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United Kingdom (11):
  - Novartis Investigative Site, Epping, Essex
  - Novartis Investigative Site, Inverness, Invernesshire
  - Novartis Investigative Site, Ipswich, Suffolk
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Denbighshire
  - Novartis Investigative Site, East Kilbride
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Portsmouth

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-seven patients were screened and 52 patients were enrolled.
Groups:
- Everolimus and Exemestane: Postmenopausal women diagnosed with oestrogen receptor positive locally advanced or metastatic breast cancer will receive everolimus at a dose of 10mg daily p.o. and exemestane 25mg daily p.o.
Period: Overall Study
Arm/Group | Everolimus and Exemestane
Started | 52
Full Analysis Set (FAS) | 49 (≥ 1 dose study drug)
Safety Analysis Set (SAF) | 49 (≥ 1 dose study drug +1 post baseline safety assessment)
Completed | 9
Not Completed | 43
Not completed — Disease progression | 26
Not completed — Adverse Event | 8
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Not completed — >1 dose of study drug | 3

BASELINE CHARACTERISTICS:
Population: FAS
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 48
  Other | 1
Weight [Mean (Standard Deviation); unit: kg] | 71.1 (15.44)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response of Everolimus and Exemestane Treatment in Postmenopausal Women With Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer
Description: The best Overall Response (OR) for each patient is determined from the sequence of investigator overall lesion responses according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1.). To be assigned a best OR of Complete Responese (CR) at least two determinations of CR at least 4 weeks apart before progression are required. To be assigned a best OR of Partial Response (PR) at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) are required.The Overall Response Rate (ORR) was defined as the proportion of patients with a best OR of confirmed CR or PR by week 48.
Time Frame: At 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
participants
  Patients with measurable disease at baseline | 39
  Patients with non-measurable disease at baseline | 10
  Best at WK 48 - Complete Response (CR) | 0
  Best at WK 48 - Partial Response (PR) | 7
  Best at WK 48 - Stable Disease (SD) | 18
  Best at WK 48 - Progressive Disease (PD) | 15
  Unknown | 1
  Missing | 8

2. Primary Outcome: Overall Response Rate of Everolimus and Exemestane Treatment in Postmenopausal Women With Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer
Description: The Overall Response Rate (ORR) was defined as the proportion of patients with a best OR of confirmed CR or PR by week 48. Treatment success is defined as: The best Overall Response (OR) for each patient is determined from the sequence of investigator overall lesion responses according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1.). To be assigned a best OR of Complete Responese (CR) at least two determinations of CR at least 4 weeks apart before progression are required. To be assigned a best OR of Partial Response (PR) at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR) are required.
Time Frame: At 48 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
Percentage of participants | 14.3 [6.0 to 27.0]

3. Secondary Outcome: Progression-free Survival (PFS) Events as Per Investigators - FAS
Description: Progression-free survival (PFS) is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment. Tumor assessment and response was evaluated according to RECIST v1.1Response was assessed by local radiology review.
Time Frame: Start of treatment to the date of event defined as first documented progression due to any cause up to approximately 48 weeks
Population: Full analysis set
Measure: Number; unit: Number of events
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
Number of events
  Deaths | 8 [12.71 to 34.29]
  Progression of disease | 25
  Number of censored observations | 16

4. Secondary Outcome: Progression-free Survival (PFS) by Median Time in Weeks as Per Investigators - FAS
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
weeks | 23.6 [12.71 to 34.29]

5. Secondary Outcome: Progression-free Survival (PFS) - % Event-free Probability Estimate - FAS
Description: Progression-free survival (PFS) is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment. Tumor assessment and response was evaluated according to RECIST v1.1Response was assessed by local radiology review. The PFS was analyzed using the Kaplan Meier method.
Time Frame: as for outcome 3
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
Percentage of participants
  Event free at 12 weeks | 67.9 [51.82 to 79.56]
  Event free at 24 weeks | 49.1 [32.98 to 63.44]
  Event free at 36 weeks | 28.9 [15.42 to 43.87]
  Event free at 48 weeks | 18.4 [7.38 to 33.19]

6. Secondary Outcome: Overall Survival (OS) Events (Number of Deaths) - FAS
Description: Overall survival (OS) is defined as the time from date of start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact. Time to median OS was not estimable.
Time Frame: Start of treatment to the date of death up to approximately 48 weeks
Population: Full analysis set
Measure: Number; unit: Number of events
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
Number of events
  Deaths | 8 [12.71 to 34.29]
  Number of censored observations | 41

7. Secondary Outcome: Overall Survival (OS) - % Event-free Probability Estimate - FAS
Description: Overall survival (OS) is defined as the time from date of start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact.
Time Frame: Start of treatment to the date of death up to approximately 48 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus and Exemestane
Number analyzed (Participants) | 49
Percentage of participants
  Event free at 12 weeks | 93.3 [80.57 to 97.78]
  Event free at 24 weeks | 83.9 [66.92 to 92.60]
  Event free at 36 weeks | 74.2 [53.02 to 86.88]
  Event free at 48 weeks | 74.2 [53.02 to 86.88]

8. Secondary Outcome: Change From Baseline EORTC Quality of Life Questionnaire of Cancer Patients QLQ-C30 at Each Time Point
Description: The QLQ-C30 is composed of multi-item scales and single-item measures including 5 functional scales, 3 symptom scales, a global health status-QoL scale, and 6 single items. Each of the multi-item scales includes a different set of items - no item occurs in more than 1 scale. High scale score=higher response level; a high score for a functional scale=a healthy level of function, high score for the global health status/QoL=high quality of life but a high score for a symptom scale / item=high level of symptomatology/problems. The principle for scoring these scales: 1.) Estimate the average of the items that contribute to the scale = raw score. 2.) Linear transformation to standardize the raw score, so that scores range from 0 to 100. Results should be interpreted with caution as the numbers of patients with available data over time were limited, and because of high variances as evidenced by large standard deviations
Time Frame: Baseline 12,24,36,48 weeks
Population: number of participants varied across visits
Measure: Mean (Standard Deviation); unit: scores
Groups:
- Week 12: Change from baseline at week 12
- Week 24: Change from baseline at Week 24
- Week 36: Change from baseline at week 36
- Week 48: Change from baseline at week 48
Arm/Group | Week 12 | Week 24 | Week 36 | Week 48
Number analyzed (Participants) | 27 | 17 | 13 | 28
scores
  Global health status/QoL: number analyzed (Participants) | 27 | 16 | 13 | 26
  Global health status/QoL | -9.0 (22.04) | -3.6 (19.71) | 1.9 (16.37) | -8.3 (22.48)
  Physical functioning | -5.1 (19.16) | -1.0 (14.52) | 4.9 (13.79) | -10.8 (29.97)
  Role functioning: number analyzed (Participants) | 26 | 16 | 12 | 27
  Role functioning | -4.5 (33.19) | 3.1 (23.74) | 8.3 (23.03) | -12.3 (30.52)
  Emotional functioning: number analyzed (Participants) | 27 | 16 | 13 | 26
  Emotional functioning | 2.6 (21.36) | -3.1 (14.87) | 7.5 (9.90) | 0.6 (21.59)
  Cognitive functioning: number analyzed (Participants) | 27 | 16 | 13 | 27
  Cognitive functioning | -8.6 (21.37) | -5.2 (17.97) | 1.3 (22.01) | -3.7 (21.35)
  Social functioning: number analyzed (Participants) | 27 | 16 | 13 | 26
  Social functioning | -9.9 (25.00) | -9.4 (24.32) | 3.8 (15.45) | -14.7 (31.74)
  Fatigue | 8.6 (26.92) | 9.5 (15.93) | 0.9 (16.64) | 7.3 (24.66)
  Nausea/ vomiting | -1.2 (15.96) | 2.9 (16.91) | -3.8 (15.45) | -2.4 (23.88)
  Pain | 1.2 (26.12) | 3.9 (24.67) | -1.3 (20.93) | 0.6 (24.64)
  Dyspnea: number analyzed (Participants) | 27 | 16 | 13 | 28
  Dyspnea | 18.5 (37.36) | 8.3 (25.82) | 2.6 (25.32) | 10.7 (27.30)
  Insomnia | 3.7 (26.69) | 2.0 (29.98) | 0 (23.57) | -3.6 (37.78)
  Appetite loss | 30.9 (40.22) | 23.5 (28.30) | 12.8 (28.99) | 16.7 (35.72)
  Constipation | 4.9 (32.95) | 11.8 (28.73) | 10.3 (21.01) | 8.3 (19.51)
  Diarrhea: number analyzed (Participants) | 27 | 16 | 13 | 27
  Diarrhea | 4.9 (25.66) | 8.3 (37.52) | -5.1 (22.96) | 7.4 (28.24)
  Financial problems: number analyzed (Participants) | 27 | 16 | 13 | 26
  Financial problems | -1.2 (21.64) | -10.4 (26.44) | -10.3 (21.01) | -2.6 (18.67)

9. Secondary Outcome: Percentage of Patient Responses in EuroQoL 5-dimension Questionnaire - FAS
Description: EuroQoL Quality of Life Scale (EQ-5D) is a standardized instrument to assess health state values is a standardized instrument to assess health state values. The EQ-5D essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The EQ-5D descriptive system is comprised of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Percentage of participants' responses were presented by visits. Results should be interpreted with caution as the numbers of patients with available data over time were limited.
Time Frame: Baseline 12,24,36,48 weeks
Measure: Number; unit: Percentage of participants
Groups:
- Day 1: Baseline
Arm/Group | Day 1 | Week 12 | Week 24 | Week 36 | Week 48
Number analyzed (Participants) | 49 | 49 | 49 | 49 | 49
Percentage of participants
  Mobility-no problem | 38.8 | 20.4 | 18.4 | 14.3 | 16.3
  Mobility-slight problem | 18.4 | 14.3 | 10.2 | 8.2 | 16.3
  Mobility-moderate problem | 32.7 | 20.4 | 8.2 | 2.0 | 14.3
  Mobility-severe problem | 6.1 | 2.0 | 0 | 2.0 | 6.1
  Mobility-unable to walk | 0 | 0 | 0 | 0 | 4.1
  Self-care - no problem | 69.4 | 44.9 | 34.7 | 24.5 | 40.8
  Self-care - slight problem | 18.4 | 4.1 | 0 | 0 | 10.2
  Self-care - moderate problem | 6.1 | 8.2 | 2.0 | 2.0 | 4.1
  Self-care -severe problem | 2.0 | 0 | 0 | 0 | 2.0
  Self-care - unable | 0 | 0 | 0 | 0 | 0
  Usual activities - no problems | 30.6 | 14.3 | 22.4 | 14.3 | 18.4
  Usual activities - slight problems | 22.4 | 16.3 | 2.0 | 8.2 | 14.3
  Usual activities - moderate problems | 28.6 | 22.4 | 12.2 | 2.0 | 12.2
  Usual activities - severe problems | 10.2 | 4.1 | 0 | 2.0 | 6.1
  Usual activities -unable to do | 4.1 | 0 | 0 | 0 | 6.1
  Pain/discomfort - none | 20.4 | 14.3 | 10.2 | 12.2 | 18.4
  Pain/discomfort - slight | 30.6 | 16.3 | 18.4 | 8.2 | 20.4
  Pain/discomfort - moderate | 40.8 | 22.4 | 8.2 | 6.1 | 14.3
  Pain/discomfort - severe | 4.1 | 4.1 | 0 | 0 | 4.1
  Pain/discomfort - extreme | 0 | 0 | 0 | 0 | 0
  Anxiety/depression - none | 44.9 | 22.4 | 18.4 | 16.3 | 22.4
  Anxiety/depression - slight | 34.7 | 22.4 | 12.2 | 10.2 | 20.4
  Anxiety/depression - moderate | 16.3 | 12.2 | 6.1 | 0 | 8.2
  Anxiety/depression - severe | 0 | 0 | 0 | 0 | 6.1
  Anxiety/depression - extreme | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in EuroQoL 5-dimension Visual Analogue Scores - FAS
Description: EuroQoL Quality of Life Scale (EQ-5D) is a standardized instrument to assess health state values. The EQ-5D essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (VAS). For the visual analogue scale, participants draw a line from a box to the point on the thermometer-like scale corresponding to their health state, 0-100 (100 = Best health state). Weights are used to score the responses to the 5 domains, with scores ranging from 0 to 1 (where a score of 1 represents a perfect state). Scores for the visual analogue scale reflect the position where participant's line crosses the thermometer-like scale. Results should be interpreted with caution as the numbers of patients with available data over time were limited, and because of high variances as evidenced by large standard deviations
Time Frame: Baseline 12,24,36,48 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 12 | Week 24 | Week 36 | Week 48
Number analyzed (Participants) | 25 | 16 | 12 | 27
units on a scale | -7.9 (18.98) | -6.1 (12.47) | -6.3 (10.03) | -11.6 (22.58)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from the First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Description: Consistent with EudracCT disclosure specifications, Novartis has reported under the Serious adverse events field "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Groups:
- Everolimus + Exemestane: Everolimus + Exemestane
Arm/Group | Everolimus + Exemestane
Serious Adverse Events (participants affected / at risk) | 22/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane (N=49)
Anaemia (Blood and lymphatic system disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Mucosal inflammation (General disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane (N=49)
Anaemia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 22
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 5
Mouth ulceration (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 8
Axillary pain (General disorders) | 4
Fatigue (General disorders) | 22
Mucosal inflammation (General disorders) | 17
Oedema peripheral (General disorders) | 3
Peripheral swelling (General disorders) | 3
Lower respiratory tract infection (Infections and infestations) | 4
Oral candidiasis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood cholesterol increased (Investigations) | 3
Blood creatinine increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 6
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 16
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 3
Depressed mood (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 18
Lymphoedema (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.